CLINICAL TRIAL: NCT02865161
Title: Open-label, Multicenter, Observational (Non-interventional) Study of Efficacy and Tolerability of Amtolmetin GuAcil in Subjects With Knee osTeoArthrosis With Dyspepsia. (AGATA)
Brief Title: Amtolmetin Gaucil in Knee Osteoarthritis
Acronym: AGATA
Status: Completed | Type: Observational
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: NISELAT-AGATA 2014
Record Dates: First submitted 2016-08-11; First posted 2016-08-12 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NISELAT: Amtolmetin guacil should be taken in fasting conditions. The recommended dose is 600 mg b.i.d. Maximum daily dose - 1800 mg
  Interventions: Drug: NISELAT

INTERVENTIONS:
Drug: NISELAT — NISELAT 600MG BD
  Other Names: AMTOLMETIN GAUCIL

SUMMARY:
This study is conducted to study the efficacy and safety of Niselat in patients with osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis is the most common rheumatic disease. Knee OA (KOA), gonarthrosis (GA), is characterized by high prevalence, progressive course with early disability of the subject, persistent pain syndrome for the treatment of which non-steroidal anti inflammatory drugs (NSAIDs) are actively used in clinical practice. It was revealed that NSAIDs may cause gastrointestinal adverse effects (AEs), from mild dyspepsia to bleeding and perforation as well as cardiovascular effects. Gastroprotection with misoprosol, Н2-receptor antagonists and proton pump inhibitors (PPI) is not always effective. NSAIDs with the lowest gastrointestinal toxicity with efficacy adequate to suppress joint pain is justified and reasonable.

Amtolmetin guacil (AMG) is a new NSAID which proved to be the least gastrointestinally toxic in experimental studies in vivo, in vitro and in comparative clinical studies. AMG does not have selectivity towards COX-2 or NO. AMG exerts gastroprotective effect due to stimulation of capsaicin receptors (vanilloid receptors) in gastrointestinal wall. To assess tolerability of amtolmetin guacil, it is first necessary to obtain data on potential reduction of dyspeptic symptoms including in subjects with these signs of NSAIDs intolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form for participation in the study;
2. KOA (based on ACR, 1987)
3. Age between 30-60 years old
4. Previous regular administration of NSAIDs for at least 4 weeks (at maximum therapeutic dose)
5. Dyspeptic symptoms (according to SODA questionnaire)
6. Pain intensity in the investigated knee joint ≥ 40 mm according to VAS
7. Subjects with systolic blood pressure ≤ 140 mm Hg and diastolic BP ≤90 mmHg against stable antihypertensive therapy.

Exclusion Criteria:

1. Contraindications to amtolmetin guacil (according to patient information leaflet)
2. Subjects with SBP ≥140 mm Hg and DBP ≥90 mm Hg
3. Signs of renal or hepatic failure;
4. Pregnancy, lactation or planning for pregnancy.
5. One of the following changes in laboratory values at screening HGB, WBC, ESR, ALT, AST.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with knee osteoarthrosis (KOA)
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Reduction in WOMAC score from baseline | Baseline to 4 weeks
  Reduced WOMAC (according to pain, rigidity and function scales) by > 20 % vs. baseline.

SECONDARY OUTCOMES:
Change in VAS | Baseline to 45 weeks
SODA Questionnaire | Baseline to 4weeks
No of adverse events | Baseline to 4 week
  Total number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Denisov L Nikolaevich, MD, Principal Investigator — Moscow, Federal State Budget Scientific Institution "Scientific Research Institute of Rheumatology named VA Nasonova"

IPD SHARING:
Plan to Share IPD: Undecided
Under review